CLINICAL TRIAL: NCT03322098
Title: Effect of Atropine or Glycopyrrolate on the Prevention of Bradycardia During Sedation Using Dexmedetomidine in Geriatric Patients Undergoing Total Knee Replacement Under Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2013-0762
Record Dates: First submitted 2017-10-23; First posted 2017-10-26 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Spinal Anesthesia
Keywords: Atropine; glycopyrrolate; bradycardia; dexmedetomidine; spinal anesthesia
MeSH Terms: conditions — Bradycardia | interventions — Atropine; Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atropine group (Active Comparator): Patients that receive atropine 0.01 mg/kg (max 0.5mg) before spinal anesthesia
  Interventions: Drug: Atropine
- Glycopyrrolate group (Active Comparator): Patients that receive glycopyrrolate 0.004mg/kg (max 0.2 mg) before spinal anesthesia
  Interventions: Drug: Glycopyrrolate

INTERVENTIONS:
Drug: Atropine — Atropine injection (0.01 mg/kg, max 0.5 mg) within 3 minutes before spinal anesthesia
  Arms: Atropine group
Drug: Glycopyrrolate — Glycopyrrolate (0.00 4mg/kg, max 0.2 mg) within 3 minutes before spinal anesthesia
  Arms: Glycopyrrolate group

SUMMARY:
Patients undergoing total knee arthroplasty with spinal anesthesia are often sedated to reduce patient discomfort due to large noises during surgery and also to reduce anxiety. Most commonly used sedatives include propofol and midazolam, but these agents often cause hypotension or respiratory depression, especially in elderly patients. Dexmedetomidine is a selective alpha 2 adrenergic drug, which acts as a sedative and also has analgesia effects. In contrast to propofol or midazolam, dexmedetomidine rarely causes respiratory depression, and therefore is often used in critically ill patients in the ICU and also in patients undergoing simple procedures. Hemodynamically, dexmedetomidine evokes a biphasic blood pressure response with a short hypertensive phase and subsequent hypotension. Bradycardia is also observed in many patients, which may lead to more serious outcomes in elderly patients who often have multiple comorbidities. Therefore, drugs to prevent bradycardia during dexmedetomidine infusion may help patients maintain a more stable hemodynamic state. The present study aims to compare the ability of atropine and glycopyrrolate to prevent bradycardia during dexmedetomidine infusion in elderly patients undergoing knee surgery with spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 65 years or older undergoing total knee replacement surgery under spinal anesthesia.
2. ASA class 1-3

Exclusion Criteria:

1. Patients with coagulation abnormalities
2. End organ diseases of liver, lung or kidney
3. Severe aortic stenosis
4. High degree AV block
5. Heart failure
6. Patients on MAO inhibitors
7. History of seizures or epilepsy
8. Glaucoma

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Pulse rate | From 5 minutes before spinal anesthesia~end of surgery (Intraoperatively)
  Measured as beats per minute, heart rate below 50 bpm or decrease of more than 30% from baseline is defined as bradycardia.
blood pressure | From 5 minutes before spinal anesthesia~end of surgery (Intraoperatively)
  Measured as mmHg, systolic blood pressure lower than 90 mmHg or decrease of more than 30% from baseline is defined as hypotension.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No